CLINICAL TRIAL: NCT04489108
Title: Tranexamic Acid for Acute Upper Gastrointestinal Bleed in Cirrhosis - A Randomized Placebo Controlled Trial
Brief Title: Tranexamic Acid for Acute Upper Gastrointestinal Bleed in Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-34
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid with Standard Medical Treatment (Experimental): Arm A will Tranexamic Acid 1g iv bolus as loading dose followed by 3g Tranexamic Acid infused over next 24 hours along with standard medical and interventional (Endoscopy) therapy.
  Interventions: Drug: Tranexamic acid; Other: Standard Medical Treatment
- Placebo + Standard Medical treatment (Active Comparator): Arm B will receive similar volume of isotonic solution (saline) along with standard medical and interventional (Endoscopy) therapy.
  Interventions: Other: Standard Medical Treatment; Other: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Tranexamic Acid 1g iv bolus as loading dose followed by 3g Tranexamic Acid infused over next 24 hours
  Arms: Tranexamic Acid with Standard Medical Treatment
Other: Standard Medical Treatment — Standard Medical Treatment
Other: Placebo — isotonic solution (saline)
  Arms: Placebo + Standard Medical treatment

SUMMARY:
The management of acute upper gastrointestinal bleeding (UGIB) is challenging in patients with cirrhosis, as it is responsible for severe complications and high mortality rates. Fibrinolytic activity of the epithelial surfaces and of the submucosal blood vessels may interfere with hematemesis and even delay healing of ulcers. Tranexamic acid (TXA) may help control the bleeding by counterbalancing cirrhosis-related hyperfibrinolysis. Still, there is a lack of unbiased data to conclude on its efficacy. Tranexamic Acid in patients with acute Upper Gastrointestinal bleed have been shown to prevent re bleed in few studies when combined with standard medical management (which generally comprises of initial fluid resuscitation, intravenous PPI , splanchnic vasoconstrictors, blood transfusions and coagulopathy corrections as per lab parameters) but no randomized placebo controlled trial has been done. The aim of this study is to evaluate the efficacy of TXA in the early treatment of acute UGIB as compared to placebo in patients with cirrhosis.

DETAILED DESCRIPTION:
Aim and Objective - AIM- To compare the efficacy and safety of tranexamic acid in reducing 5-day treatment failure (i.e., failure to control bleed) in patients with cirrhosis presenting with Upper GI bleed

Primary Objective:

Proportion of patients developing five-day treatment failure (i.e., failure to control bleed)

Secondary Objectives:

1. Failure to prevent rebleed within 6 weeks
2. Clinically significant rebleed within 6 weeks (monitored by hemoglobin drop by 3g/dl, need of blood transfusion)
3. Need for salvage therapy (tamponade, additional endoscopic therapy, TIPS, surgery etc.)
4. Blood product and component requirements
5. Days of ICU/hospital stay
6. Thromboembolic events (deep vein thrombosis, pulmonary embolism, stroke, myocardial infarction etc)
7. Other complications post bleed (including other significant cardiac event, sepsis, pneumonia, respiratory failure, Acute Kidney Injury, seizures etc)
8. Mortality attributed to failure to control bleed.

Methodology:

* Study population: Patients of Cirrhosis presenting with Acute Upper Gastrointestinal bleed
* Study design:Single Centre, Double Blinded (Patient and Treating physician), Placebo Controlled (Saline), Randomised Controlled Trial
* Study period: 1.5 years from the date of ethics approval

Sample size with justification:

- Assuming 5-day treatment failure in Placebo arm around 25% and 15 % in the treatment arm. Alpha- 5%, Power- 80%. The investigators need to enroll 542 cases with 271 in each group. Further assuming 10% dropout, it is decided to enroll 600 cases , randomly allocated into two arms by Block Randomization with Block size of 10. An interim analysis will be done at reaching total of 300 sample size.

Intervention:

- Patients will be randomized into two Arms A & B. Both the patient and treating physician are blinded Arm A- Tranexamic Acid arm- Will receive Tranexamic Acid 1g iv bolus as loading dose followed by 3g Tranexamic Acid infused over next 24 hours along with standard medical and interventional (Endoscopy) therapy.

Arm B- Will receive similar volume of isotonic solution (saline) along with standard medical and interventional (Endoscopy) therapy.

Monitoring and Assessment:

1. Five-day treatment failure (i.e., failure to control bleed)- defined as death or need to change therapy defined by one of the following criteria:

   * fresh hematemesis or
   * nasogastric aspiration of ≥100 mL of fresh blood ≥2 hours after the start of a specific drug treatment or
   * therapeutic endoscopy;
   * development of hypovolaemic shock;
   * 3 g drop in hemoglobin (Hb) (9% drop of hematocrit) within any 24-hour period if no transfusion is administered.
2. Failure to prevent rebleeding defined as a single episode of clinically significant rebleeding after day 5 until 6 weeks, and
3. Clinically significant rebleeding defined as recurrent melena or hematemesis resulting in any of the following after day 5 until 6 weeks:

   * hospital admission,
   * blood transfusion,
   * 3 g drop in haemoglobin, or
   * Death

Other treatments given

1. Conditioning (intravenous access, tracheal intubation or other airways management technique if needed)
2. Medical interventions (immediate splanchnic vasopressors: terlipressin or somatostatin and derivatives before endoscopy (up to 5 days)
3. PPIs in case of suspicion of associated peptic ulcer
4. Antibiotics during 5 days and later as needed
5. Hemodynamic stabilisation (fluid infusion, systemic vasopressors as noradrenalin or adrenalin);
6. Technical interventions (endoscopy as soon as possible, within 12 hours, and haemostatic interventions like EVL, Glue, Dannis-Ella stent, if feasible early TIPS within 72 hours (Child C or B with active bleeding at endoscopy)
7. Secondary prophylaxis (from day 6 after onset): beta blockers if stable will be mandatory for the secondary prophylaxis.
8. ROTEM based correction will be given for patients having nonvariceal upper GI bleeding (diagnosed after doing upper GI endoscopy and showing ongoing bleed form a nonvariceal source at that time); and significant coagulopathy assessed by INR > 1.8 and/or PLTs < 50 × 109/L.

Assessment of Fibrinolysis:

1. FDP (Fibrin Degradation Products)
2. d-Dimer assay
3. Fibrinogen
4. FIBTEM-EXTEM

Data to be Collected

1. Hemogram, PT/INR, LFT, KFT (baseline, D1, 3, 5, 7, 14, 28, 42 and as needed)
2. d-Dimer, FDP, Fibrinogen, ROTEM (FIBTEM/EXTEM): (baseline, day 1, 3, 5)
3. USG with doppler SPA, AFP, sugar (F),Chest Xray other etiological investigations as needed: baseline
4. UGIE findings
5. Other clinical parameters such as CTP score, MELD score, Heart rate, Blood Pressure

ELIGIBILITY:
Inclusion Criteria:

1. Patients greater than 18 years of age
2. Presenting with Acute UGI bleed (< 24hrs from onset).
3. Cirrhosis (Known Or suspected on clinical, biological, radiological data or the patient's history) with CTP B / C (i.e. CTP >/=7) or ACLF (with clinical evidence of cirrhosis).

Exclusion Criteria:

1. Non cirrhotic patients
2. Known allergy to Tranexamic Acid
3. Patients with clinical evidence of DIC (Disseminated Intravascular Coagulation) like coagulopathy patches/ haematuria / uncontrolled epistaxis etc.
4. Patients with Chronic Kidney Disease.
5. History of recent Cerebro Vascular Accident (CVA) [in the past 6 months] or patients with thrombotic events [Portal Vein thrombosis /Hepatic vein thrombosis /other sites thrombosis]. HCC with tumour thrombosis will be included
6. Any history of seizures, myocardial infarction
7. Pregnancy/lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients developing five-day treatment failure in both the groups | 5 day

SECONDARY OUTCOMES:
Number of patients with failure to prevent rebleed in both group | 6 weeks
Clinically significant rebleed in both groups | 6 weeks
  Clinically significant rebleed as monitored by hemoglobin drop by 3g/dl, need of blood transfusion
Number of patients who will require salvage therapy in both groups | 6 weeks
Number of patients who will require Blood product and component in both groups | 6 weeks
Number of days in Intensive Care Unit in both groups | 6 weeks
Number of days in hospital in both groups | 6 weeks
Number of patients with deep vein thrombosis in both groups | 6 weeks
Number of patients with pulmonary embolism in both groups | 6 weeks
Number of patients with stroke in both groups | 6 weeks
Number of patients with myocardial infarction in both groups | 6 weeks
Number of patients with Adverse Events associated with post bleed in both groups | 6 weeks
Number of patients with Mortality attributed to failure to control bleed in both groups | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided